CLINICAL TRIAL: NCT06777654
Title: Unilateral and Bilateral Approaches to Robotic Therapy Hybridized With Mirror Therapy in Stroke Rehabilitation
Brief Title: Robotic Therapy Hybridized With Mirror Therapy in Stroke Rehabilitation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202410139RIND
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-01

CONDITIONS: Stroke
Keywords: Robotic Rehabilitation; Mirror Therapy; Stroke Rehabilitation; Computerized Rehabilitation; Randomized Controlled Trial
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unilateral RT plus unilateral innovative MT (Experimental): Unilateral robotic therapy (RT) with computerized visual feedback plus unilateral innovative mirror therapy (MT)
  Interventions: Other: Robotic therapy (RT); Other: Mirror therapy (MT)
- Bilateral RT plus bilateral innovative MT (Experimental): Bilateral robotic therapy (RT) with computerized visual feedback plus bilateral innovative mirror therapy (MT)
  Interventions: Other: Robotic therapy (RT); Other: Mirror therapy (MT)
- Dose-matched conventional rehabilitation (Active Comparator): Dose-matched conventional rehabilitation as the control
  Interventions: Other: Dose-matched control intervention

INTERVENTIONS:
Other: Robotic therapy (RT) — The Bi-Manu-Track (BMT) robot will be provided as the robotic practice. The BMT can be switched from the bilateral practice modules involving bilateral upper limbs to the unilateral module involving the affected upper limb. According to the group assignment, participants will practice the unilateral or bilateral module of BMT training.
  Arms: Bilateral RT plus bilateral innovative MT; Unilateral RT plus unilateral innovative MT
Other: Mirror therapy (MT) — The innovative mirror therapy (MT) program will be conducted with computerized mirror visual feedback and the conventional mirror box therapy. The unilateral MT group will practice on the unilateral module, while the bilateral MT group will practice based on the bilateral module. In the unilateral module, the affected hand will be static on the knee. In contrast, during bilateral MT, participants will be asked to do the same movements using the unaffected and affected arms as symmetrically as possible.
  Arms: Bilateral RT plus bilateral innovative MT; Unilateral RT plus unilateral innovative MT
Other: Dose-matched control intervention — Participants in the control group will receive therapist-mediated rehabilitation per session.
  Arms: Dose-matched conventional rehabilitation

SUMMARY:
The goal of this clinical trial is to compare the effects of three groups: (1) unilateral robotic therapy with computerized visual feedback plus unilateral innovative mirror therapy, (2) bilateral robotic therapy with computerized visual feedback plus bilateral innovative mirror therapy, and (3) dose-matched conventional rehabilitation as the control. The investigators will also study the factors predictive of treatment success, identify key predictors of clinical improvement, and distinguish patient profiles most likely to benefit from each regimen. The findings of this clinical trial are expected to advance knowledge about the synergistic effects of unilateral and bilateral hybrid programs. The predictive study of treatment outcomes will inform patient selection in precision rehabilitation toward personalized stroke management.

ELIGIBILITY:
Inclusion Criteria:

(1) a first ever-stroke≧3 months and less than 2 years, (2) age range between 30 to 80 years, (3) baseline Fugl-Meyer Assessment-Upper Extremity subscale (FMA-UE) between 18 to 56, (4) no excessive muscle spasticity of the affected extremities (Modified Ashworth Scale < 3 at any joints), (5) able to follow examiners' commands and study instructions (Montreal Cognitive Assessment score≧22), and (6) no fracture of upper extremities within the past 3 months, and (7) no participation in any other experimental rehabilitation or drug studies during study period of this project.

Exclusion Criteria:

(1) acute inflammation and pain, (2) receiving botulinum toxin injections within the past 3 months, and (3) concomitant neurologic, neuromuscular or orthopedic conditions that may interfere with participation in this research.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment-Upper Extremity subscale (FMA-UE) | Baseline, 6 weeks, and 18 weeks

SECONDARY OUTCOMES:
Grip and pinch strength | Baseline, 6 weeks, and 18 weeks
Box and Block Test (BBT) | Baseline, 6 weeks, and 18 weeks
Revised Nottingham Sensory Assessment (rNSA) | Baseline, 6 weeks, and 18 weeks
Motor Activity Log (MAL) | Baseline, 6 weeks, and 18 weeks
ABILHAND Questionnaire | Baseline, 6 weeks, and 18 weeks
Functional Ambulation Category (FAC) | Baseline, 6 weeks, and 18 weeks
Stroke Impact Scale Version 3.0 (SIS 3.0) | Baseline, 6 weeks, and 18 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Wan Fang Hospital, Taipei Medical University, Taipei
  - National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No